CLINICAL TRIAL: NCT06537869
Title: The New Internet Generation: iCBT Treatment for Seniors With Mild-moderate Depression - a Pragmatic Randomised Controlled Trial in the Primary Care Context
Brief Title: iCBT for Seniors With Depression in Primary Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: iCBT-Senior-DEP-2024-PRCT
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Depression Mild; Depression Moderate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iCBT Senior (Experimental): iCBT depression program with minimal therapist contact offered within 14 days from inclusion and with a duration of 10-12 weeks. Contact via email or telephone every week (therapist/nurse)
  Interventions: Behavioral: iCBT for depression
- Depression treatment-as-usual Senior (Active Comparator): Depression treatment-as-usual for patient >65 years
  Interventions: Behavioral: iCBT for depression

INTERVENTIONS:
Behavioral: iCBT for depression — iCBT depression program with minimal therapist contact offered within 14 days from inclusion and with a duration of 10-12 weeks. Contact via email or telephone every week (therapist/nurse)

SUMMARY:
This clinical trial aims to evaluate the potential benefits of internet cognitive behavioural therapy (iCBT) for elderly patients with mild/moderate depression and compare its effectiveness with the current treatment as usual (TAU) at primary care centres (PCCs).

The specific aims are to study if:

iCBT is as effective as TAU in reducing depressive symptoms iCBT is as effective as TAU in increasing quality of life iCBT is as effective as TAU in increasing the function in patients >65 years and older with mild/moderate depression attending primary care, with the perspective of 36 months.

Participants will:

Work with the iCBT program (10-12 weeks) or become TAU at their PCCs. Followed-up at 3, 6, 12, 24 and 36 months of their symptoms, quality of life and function.

DETAILED DESCRIPTION:
Study Objective:

The primary aim is to determine if iCBT is as effective for treating mild-moderate depression in older adults (<65) as it is for younger age groups. The study will assess various outcomes throughout 3, 6, 12, 24, and 36 months, including depressive symptoms, quality of life, workability, relationships, activities of daily living, and social participation.

Trial Design:

It's a randomised controlled trial (RCT) with two groups: intervention (iCBT) and control (TAU). The pragmatic design closely resembles real-world primary care conditions to ensure the results apply to routine clinical practice.

Population:

Participants will be recruited from primary care centres (PCCs) in Sweden, targeting individuals over 65 years diagnosed with mild to moderate depressive symptoms. The study aims to include all eligible patients from participating PCCs, ensuring a broad representation of the target population.

Intervention and Control:

Intervention:

iCBT program with minimal therapist contact, initiated promptly after inclusion and lasting 10-12 weeks. Weekly therapist/nurse contact via email or telephone is part of the intervention.

Control:

TAU according to Swedish National Guidelines may include guided self-help, face-to-face CBT (excluding iCBT), and/or antidepressants provided by GPs or nurses at the PCCs.

Patient Selection and Randomization:

Patients will be screened using standardised guidelines (NICE guidelines for depression), diagnosed via the MINI diagnostic interview (Mini International Neuropsychiatric Interview), and randomised centrally to avoid bias. Due to the nature of the intervention, blinding at the patient level isn't feasible, but efforts will be made to blind researchers during data analysis.

Follow-up and Data Collection:

Multiple follow-up points up to 36 months will allow the researchers to assess the longer-term effects of iCBT compared to TAU. Quantitative outcomes will be supplemented by qualitative data from focus group interviews with patients and staff, exploring their experiences with iCBT.

Focus Group Interviews:

These will involve patients and staff separately, aiming to gather insights into the acceptability, feasibility, and perceived effectiveness of iCBT in a primary care setting. Qualitative analysis methods will be used to interpret and contextualise the findings from these interviews.

ELIGIBILITY:
Inclusion Criteria:

* All patients >65, attending PCCs engaged in the trial, with mood as well as somatic complaints will be asked about depressive symptoms during the last 2 weeks by NICE guidelines for depression.
* All patients diagnosed with minor/major depression and not belonging to exclusion criteria and willing to take part in the trial will be diagnosed via the Mini International Neuropsychiatric Interview (M.I.N.I.) by a psychologist/specially trained nurse and have a General Practitioner (GP) somatic consultation

Exclusion Criteria:

Patients diagnosed with:

* severe depression
* prior suicide attempt or currently at medium to high risk of suicide (MADRS-S question 9>3 points or MINI suicide >9)
* bipolar disorder
* psychosis
* addiction
* cognitive impairment
* not speaking or understanding Swedish.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
MADRS-S (Montgomery and Asberg Depression Rating Scale) | Change from baseline scores MADRS-S scale at 3 months
  What is the effect of iCBT on participants' symptoms of depression (measured as a change in score in MADRS-S from baseline to 3 months after baseline)?
  Scale:
  0 to 6 - normal/symptom absent 7 to 19 - mild depression 20 to 34 - moderate depression >34 - severe depression
MADRS-S (Montgomery and Asberg Depression Rating Scale) | Change from baseline scores MADRS-S scale at 6 months
  What is the effect of iCBT on participants' symptoms of depression (measured as a change in score in MADRS-S from baseline to 6 months after baseline)?
  Scale:
  0 to 6 - normal/symptom absent 7 to 19 - mild depression 20 to 34 - moderate depression >34 - severe depression
MADRS-S (Montgomery and Asberg Depression Rating Scale) | Change from baseline scores MADRS-S scale at 12 months
  What is the effect of iCBT on participants' symptoms of depression (measured as a change in score in MADRS-S from baseline to 12 months after baseline)?
  Scale:
  0 to 6 - normal/symptom absent 7 to 19 - mild depression 20 to 34 - moderate depression >34 - severe depression
MADRS-S (Montgomery and Asberg Depression Rating Scale) | Change from baseline scores MADRS-S scale at 24 months
  What is the effect of iCBT on participants' symptoms of depression (measured as a change in score in MADRS-S from baseline to 24 months after baseline)?
  Scale:
  0 to 6 - normal/symptom absent 7 to 19 - mild depression 20 to 34 - moderate depression >34 - severe depression
MADRS-S (Montgomery and Asberg Depression Rating Scale) | Change from baseline scores MADRS-S scale at 36 months
  What is the effect of iCBT on participants' symptoms of depression (measured as a change in score in MADRS-S from baseline to 36 months after baseline)?
  Scale:
  0 to 6 - normal/symptom absent 7 to 19 - mild depression 20 to 34 - moderate depression >34 - severe depression

SECONDARY OUTCOMES:
The 5-level EQ-5D version (EQ-5D-5L) EuroQol 5-Dimension | Change from baseline scores EQ-5D scale at 3 months
  Scale Title: EQ-5D-5L. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. 1 = no difficulties and 5 = very large difficulties. These single-digit codes can be combined into a five-digit code that corresponds to a specific health profile. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  What is the effect of iCBT on participants' health-related quality of life (measured by the change in scores in EQ-5D from baseline to 3 months after baseline)?
The 5-level EQ-5D version (EQ-5D-5L) | Change from baseline scores EQ-5D scale at 6 months
  What is the effect of iCBT on participants' health-related quality of life (measured by the change in scores in EQ-5D from baseline to 6 months after baseline? The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has five levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate their health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
The 5-level EQ-5D version (EQ-5D-5L) | Change from baseline scores EQ-5D scale at 12 months
  What is the effect of iCBT on participants' health-related quality of life (measured by the change in scores in EQ-5D from baseline to 12 months after baseline? The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has five levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate their health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
The 5-level EQ-5D version (EQ-5D-5L) | Change from baseline scores EQ-5D scale at 24 months
  What is the effect of iCBT on participants' health-related quality of life (measured by the change in scores in EQ-5D from baseline to 24 months after baseline? The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has five levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate their health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
The 5-level EQ-5D version (EQ-5D-5L) | Change from baseline scores EQ-5D scale at 36 months
  What is the effect of iCBT on participants' health-related quality of life (measured by the change in scores in EQ-5D from baseline to 36 months after baseline? The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has five levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate their health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Work ability | Change from baseline scores WAI scale at 3 months
  Scale Title: Work Ability Index (WAI) Minimum Value: 7 Maximum Value: 49 Higher Scores Mean: A better outcome. The WAI is used to assess an individual's work ability based on their health and work capacity.What is the effect of iCBT on participants' work ability (measured as change in scores in WAI from baseline to 3 months after baseline). Work ability was measured by means of the Work Ability Index (WAI) which consists in a 7-part self-assessment: current ability, work ability in relation to physical and mental demands of the job, reported diagnosed diseases, estimated impairment due to health status, sick leave over the last 12 months, self-prognosis of work ability in the 2 years to come and mental resources of the individual. The WAI measured in this way ranges from 7 to 49 points and 4 categories have been suggested to describe WAI levels: poor (7-27), moderate (28-36), good (37-43) and excellent (44-49).
Work ability | Change from base-line scores WAI scale at 6 months
  What is the effect of iCBT on participants' work ability (measured as change in scores in WAI from baseline to 6 months after baseline). Work ability was measured by means of the Work Ability Index (WAI) which consists in a 7-part self-assessment: current ability, work ability in relation to physical and mental demands of the job, reported diagnosed diseases, estimated impairment due to health status, sick leave over the last 12 months, self-prognosis of work ability in the 2 years to come and mental resources of the individual. The WAI measured in this way ranges from 7 to 49 points and 4 categories have been suggested to describe WAI levels: poor (7-27), moderate (28-36), good (37-43) and excellent (44-49).
Work ability | Change from base-line scores WAI scale at 12 months
  What is the effect of iCBT on participants' work ability (measured as change in scores in WAI from baseline to 12 months after baseline). Work ability was measured by means of the Work Ability Index (WAI) which consists in a 7-part self-assessment: current ability, work ability in relation to physical and mental demands of the job, reported diagnosed diseases, estimated impairment due to health status, sick leave over the last 12 months, self-prognosis of work ability in the 2 years to come and mental resources of the individual. The WAI measured in this way ranges from 7 to 49 points and 4 categories have been suggested to describe WAI levels: poor (7-27), moderate (28-36), good (37-43) and excellent (44-49).
Work ability | Change from base-line scores WAI scale at 24 months
  What is the effect of iCBT on participants' work ability (measured as change in scores in WAI from baseline to 24 months after baseline). Work ability was measured by means of the Work Ability Index (WAI) which consists in a 7-part self-assessment: current ability, work ability in relation to physical and mental demands of the job, reported diagnosed diseases, estimated impairment due to health status, sick leave over the last 12 months, self-prognosis of work ability in the 2 years to come and mental resources of the individual. The WAI measured in this way ranges from 7 to 49 points and 4 categories have been suggested to describe WAI levels: poor (7-27), moderate (28-36), good (37-43) and excellent (44-49).
Work ability | Change from base-line scores WAI scale at 36 months
  What is the effect of iCBT on participants' work ability (measured as change in scores in WAI from baseline to 36 months after baseline). Work ability was measured by means of the Work Ability Index (WAI) which consists in a 7-part self-assessment: current ability, work ability in relation to physical and mental demands of the job, reported diagnosed diseases, estimated impairment due to health status, sick leave over the last 12 months, self-prognosis of work ability in the 2 years to come and mental resources of the individual. The WAI measured in this way ranges from 7 to 49 points and 4 categories have been suggested to describe WAI levels: poor (7-27), moderate (28-36), good (37-43) and excellent (44-49).
WHODAS 12 2.0 (WORLD HEALTH ORGANIZATION DISABILITY ASSESSMENT SCHEDULE 2.0), 12-item version, self-administered | Change from base-line scores WHODAS scale at 3 months
  What is the effect of iCBT on participants' disability work (measured as a change in scores in WHODAS from baseline to 3 months after baseline)? This questionnaire asks about difficulties due to health conditions. Health conditions include diseases or illnesses, other health problems that may be short or long-lasting, injuries, mental or emotional problems, and problems with alcohol or drugs.
  Review the past 30 days and answer these questions, thinking about how difficult participant had to do the following activities. WHODAS 2.0 covers 6 Domains of Functioning, including Cognition - understanding & communicating; mobility- moving & getting around; self-care- hygiene, dressing, eating & staying alone; getting along- interacting with other people; life activities- domestic responsibilities, leisure, work & school, Participation- joining in community activities
WHODAS 12 2.0 (WORLD HEALTH ORGANIZATION DISABILITY ASSESSMENT SCHEDULE 2.0), 12-item version, self-administered | Change from base-line scores WHODAS scale at 6 months
  What is the effect of iCBT on participants' disability work (measured as a change in scores in WHODAS from baseline to 6 months after baseline)? This questionnaire asks about difficulties due to health conditions. Health conditions include diseases or illnesses, other health problems that may be short or long-lasting, injuries, mental or emotional problems, and problems with alcohol or drugs.
  Review the past 30 days and answer these questions, thinking about how difficult participant had to do the following activities. WHODAS 2.0 covers 6 Domains of Functioning, including Cognition - understanding & communicating; mobility- moving & getting around; self-care- hygiene, dressing, eating & staying alone; getting along- interacting with other people; life activities- domestic responsibilities, leisure, work & school, Participation- joining in community activities
WHODAS 12 2.0 (WORLD HEALTH ORGANIZATION DISABILITY ASSESSMENT SCHEDULE 2.0), 12-item version, self-administered | Change from base-line scores WHODAS scale at 12 months
  What is the effect of iCBT on participants' disability work (measured as a change in scores in WHODAS from baseline to 12 months after baseline)? This questionnaire asks about difficulties due to health conditions. Health conditions include diseases or illnesses, other health problems that may be short or long-lasting, injuries, mental or emotional problems, and problems with alcohol or drugs.
  Review the past 30 days and answer these questions, thinking about how difficult participant had to do the following activities. WHODAS 2.0 covers 6 Domains of Functioning, including Cognition - understanding & communicating; mobility- moving & getting around; self-care- hygiene, dressing, eating & staying alone; getting along- interacting with other people; life activities- domestic responsibilities, leisure, work & school, Participation- joining in community activities
WHODAS 12 2.0 (WORLD HEALTH ORGANIZATION DISABILITY ASSESSMENT SCHEDULE 2.0), 12-item version, self-administered | Change from base-line scores WHODAS scale at 24 months
  What is the effect of iCBT on participants' disability work (measured as a change in scores in WHODAS from baseline to 24 months after baseline)? This questionnaire asks about difficulties due to health conditions. Health conditions include diseases or illnesses, other health problems that may be short or long-lasting, injuries, mental or emotional problems, and problems with alcohol or drugs.
  Review the past 30 days and answer these questions, thinking about how difficult participant had to do the following activities. WHODAS 2.0 covers 6 Domains of Functioning, including Cognition - understanding & communicating; mobility- moving & getting around; self-care- hygiene, dressing, eating & staying alone; getting along- interacting with other people; life activities- domestic responsibilities, leisure, work & school, Participation- joining in community activities
WHODAS 12 2.0 (WORLD HEALTH ORGANIZATION DISABILITY ASSESSMENT SCHEDULE 2.0), 12-item version, self-administered | Change from base-line scores WHODAS scale at 36 months
  What is the effect of iCBT on participants' disability work (measured as a change in scores in WHODAS from baseline to 36 months after baseline)? This questionnaire asks about difficulties due to health conditions. Health conditions include diseases or illnesses, other health problems that may be short or long-lasting, injuries, mental or emotional problems, and problems with alcohol or drugs.
  Review the past 30 days and answer these questions, thinking about how difficult participant had to do the following activities. WHODAS 2.0 covers 6 Domains of Functioning, including Cognition - understanding & communicating; mobility- moving & getting around; self-care- hygiene, dressing, eating & staying alone; getting along- interacting with other people; life activities- domestic responsibilities, leisure, work & school, Participation- joining in community activities
Use of Antidepressants | Antidepressant use will be assessed at baseline and after 12 months of participation in the study.
  The use of antidepressants will be assessed as a secondary outcome measure in this study to understand its impact on the treatment of mild to moderate depression in individuals aged 66 and above. Antidepressant use will be compared between the intervention group (receiving iCBT) and the control group (receiving Treatment-As-Usual, TAU) over a 12-month period.
General Self-Efficacy Scale (GSE) | Change from base-line scores GSE scale at 3 months
  The General Self-Efficacy Scale is correlated to emotion, optimism, work, satisfaction. Negative coefficients were found for depression, stress, health complaints, burnout, and anxiety. Scoring: Not at all true, Hardly true, Moderately true, Exactly true, All questions 1 2 3 4. The total score is calculated by finding the sum of the all items. For the GSE, the total score ranges between 10 and 40, with a higher score indicating more self-efficacy.
General Self-Efficacy Scale (GSE) | Change from base-line scores GSE scale at 6 months
  The General Self-Efficacy Scale is correlated to emotion, optimism, work, satisfaction. Negative coefficients were found for depression, stress, health complaints, burnout, and anxiety. Scoring: Not at all true, Hardly true, Moderately true, Exactly true, All questions 1 2 3 4. The total score is calculated by finding the sum of the all items. For the GSE, the total score ranges between 10 and 40, with a higher score indicating more self-efficacy.
General Self-Efficacy Scale (GSE) | Change from base-line scores GSE scale at 12 months
  The General Self-Efficacy Scale is correlated to emotion, optimism, work, satisfaction. Negative coefficients were found for depression, stress, health complaints, burnout, and anxiety. Scoring: Not at all true, Hardly true, Moderately true, Exactly true, All questions 1 2 3 4. The total score is calculated by finding the sum of the all items. For the GSE, the total score ranges between 10 and 40, with a higher score indicating more self-efficacy.
General Self-Efficacy Scale (GSE) | Change from base-line scores GSE scale at 24 months
  The General Self-Efficacy Scale is correlated to emotion, optimism, work, satisfaction. Negative coefficients were found for depression, stress, health complaints, burnout, and anxiety. Scoring: Not at all true, Hardly true, Moderately true, Exactly true, All questions 1 2 3 4. The total score is calculated by finding the sum of the all items. For the GSE, the total score ranges between 10 and 40, with a higher score indicating more self-efficacy.
General Self-Efficacy Scale (GSE) | Change from base-line scores GSE scale at 36 months
  The General Self-Efficacy Scale is correlated to emotion, optimism, work, satisfaction. Negative coefficients were found for depression, stress, health complaints, burnout, and anxiety. Scoring: Not at all true, Hardly true, Moderately true, Exactly true, All questions 1 2 3 4. The total score is calculated by finding the sum of the all items. For the GSE, the total score ranges between 10 and 40, with a higher score indicating more self-efficacy.
The Health Literacy Survey European Questionnaire (HLS-EU-Q16) | Change from base-line scores HLSE-EU-Q16 scale at 3 months
  The HLS-EU-Q16, or the Health Literacy Survey European Questionnaire (short version with 16 questions), is a standardized tool designed to measure health literacy in populations. Health literacy refers to an individual's ability to access, understand, appraise, and apply information to make informed decisions regarding their health. Each question in the HLS-EU-Q16 is answered on a Likert scale with four response options: Very difficult (1 point), Fairly difficult (2 points), Fairly easy (3 points), Very easy (4 points). To calculate the total score, sum the points for all 16 questions. The total score can range from 16 to 64 points. Low points are Inadequate Health Literacy.
The Health Literacy Survey European Questionnaire (HLS-EU-Q16) | Change from base-line scores HLSE-EU-Q16 scale at 6 months
  The HLS-EU-Q16, or the Health Literacy Survey European Questionnaire (short version with 16 questions), is a standardized tool designed to measure health literacy in populations. Health literacy refers to an individual's ability to access, understand, appraise, and apply information to make informed decisions regarding their health. Each question in the HLS-EU-Q16 is answered on a Likert scale with four response options: Very difficult (1 point), Fairly difficult (2 points), Fairly easy (3 points), Very easy (4 points). To calculate the total score, sum the points for all 16 questions. The total score can range from 16 to 64 points. Low points are Inadequate Health Literacy.
The Health Literacy Survey European Questionnaire (HLS-EU-Q16) | Change from base-line scores HLSE-EU-Q16 scale at 12 months
  The HLS-EU-Q16, or the Health Literacy Survey European Questionnaire (short version with 16 questions), is a standardized tool designed to measure health literacy in populations. Health literacy refers to an individual's ability to access, understand, appraise, and apply information to make informed decisions regarding their health. Each question in the HLS-EU-Q16 is answered on a Likert scale with four response options: Very difficult (1 point), Fairly difficult (2 points), Fairly easy (3 points), Very easy (4 points). To calculate the total score, sum the points for all 16 questions. The total score can range from 16 to 64 points. Low points are Inadequate Health Literacy.
The Health Literacy Survey European Questionnaire (HLS-EU-Q16) | Change from base-line scores HLSE-EU-Q16 scale at 24 months
  The HLS-EU-Q16, or the Health Literacy Survey European Questionnaire (short version with 16 questions), is a standardized tool designed to measure health literacy in populations. Health literacy refers to an individual's ability to access, understand, appraise, and apply information to make informed decisions regarding their health. Each question in the HLS-EU-Q16 is answered on a Likert scale with four response options: Very difficult (1 point), Fairly difficult (2 points), Fairly easy (3 points), Very easy (4 points). To calculate the total score, sum the points for all 16 questions. The total score can range from 16 to 64 points. Low points are Inadequate Health Literacy.
The Health Literacy Survey European Questionnaire (HLS-EU-Q16) | Change from base-line scores HLSE-EU-Q16 scale at 36 months
  The HLS-EU-Q16, or the Health Literacy Survey European Questionnaire (short version with 16 questions), is a standardized tool designed to measure health literacy in populations. Health literacy refers to an individual's ability to access, understand, appraise, and apply information to make informed decisions regarding their health. Each question in the HLS-EU-Q16 is answered on a Likert scale with four response options: Very difficult (1 point), Fairly difficult (2 points), Fairly easy (3 points), Very easy (4 points). To calculate the total score, sum the points for all 16 questions. The total score can range from 16 to 64 points. Low points are Inadequate Health Literacy.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Hange, Ass Prof, Principal Investigator — Göteborg University
Locations (1):
- University of Gothenburg, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-08-15): https://cdn.clinicaltrials.gov/large-docs/69/NCT06537869/SAP_000.pdf